CLINICAL TRIAL: NCT06474598
Title: A Open Label, Parallel Group Phase IIA, Adaptive Design Study of MTX228 in Adult Subjects With Type 1 Diabetes and Preserved β-Cell Function
Brief Title: An Adaptive Design Study of MTX228
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTX228-2024
Record Dates: First submitted 2024-04-08; First posted 2024-06-25 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 100 mg QD (Active Comparator): Participants will be assigned to receive 3 months oral tablet administration of MTX228 at the 100mg QD dose
  Interventions: Drug: MTX228; Device: DEXCOM G6
- 100 mg BID (Active Comparator): Participants will be assigned to receive 3 months oral tablet administration of MTX228 at the 100mg BID dose
  Interventions: Drug: MTX228; Device: DEXCOM G6
- 200 mg QD (Active Comparator): Participants will be assigned to receive 3 months oral tablet administration of MTX228 at the 200mg BID dose
  Interventions: Drug: MTX228; Device: DEXCOM G6

INTERVENTIONS:
Drug: MTX228 — Tolimidone was developed as a treatment for gastric ulcers but did not advance beyond phase 2 clinical trials because of lack of efficacy. Subsequently, tolimidone has been identified as an activator of Lyn kinase and was considered as a treatment for type 2 diabetes as an insulin sensitizer because of Lyn's interaction with insulin signaling molecules. More recently, Lyn has been identified as a critical regulator of beta-cell mass, with genetic and biochemical inactivation of Lyn provoking beta-cell death in isolated human islets and precipitated diabetes in mice, and activation of Lyn stimulating beta-cell survival and beta-cell proliferation. These findings strongly suggest that small molecule activators of Lyn, such as Tolimidone, could represent new therapeutic options to promote beta-cell regeneration in type 1 diabete
  Other Names: Tolimidone
Device: DEXCOM G6 — To monitor participants blood glucose levels continuously

SUMMARY:
MTX228 has been identified as a medication that might allow the re-growth of insulin producing beta cells in people with Type 1 Diabetes. Promoting the re-growth of lost beta cells would be beneficial to people with Type 1 Diabetes because it would allow them to take less insulin by injection and would improve their overall blood sugar control while reducing the risk and rate of low blood sugars. This open-label dose selection study aims to determine the optimal dose ofMTX228 for use in a future phase IIb study.

The purpose is to investigate the relative effectiveness of different doses of MTX228 and to select the most effective dose for further investigation in a phase 2b study.

DETAILED DESCRIPTION:
MTX228 was developed as a treatment for gastric ulcers but did not advance beyond phase 2 clinical trials because of lack of efficacy. Subsequently, MTX228 has been identified as an activator of Lyn kinase and was considered as a treatment for type 2 diabetes as an insulin sensitizer because of Lyn's interaction with insulin signaling molecules. More recently, Lyn has been identified as a critical regulator of beta-cell mass, with genetic and biochemical inactivation of Lyn provoking beta-cell death in isolated human islets and precipitated diabetes in mice, and activation of Lyn stimulating beta-cell survival and beta-cell proliferation. These findings strongly suggest that small molecule activators of Lyn, such as MTX228, could represent new therapeutic options to promote beta-cell regeneration in type 1 diabetes.

MTX228 has not been testing in clinical studies in type 1 diabetes and the optimal dose to use is not clear from the clinical trial in type 2 diabetes, where lower doses (100 mg once or twice daily) were more effective than higher doses (200 mg once or twice daily). The purpose of this study is to compare the effect of different doses of MTX228 in order to determine the most effective dose to move forward in a subsequent phase 2b study.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of T1DM with onset before the age of 35 requiring continuous treatment with insulin within 1 year of diagnosis and the presence of positive T1DM autoantibody titer if diagnosed after age 35 (past or present
* HbA1c between 6.0 - 10.0 %.
* Willing to wear study-provided CGM and share CGM data via cloud.
* Diagnosis of T1DM ≥1year at time of screening.
* Fasting or random (post-prandial) C-peptide level ≥ 100 pmol/l (or 0.3 ng/mL) during screening or pre-screening. Pre-screening C-peptide levels may be obtained by the study team (subject to patient's written consent) up to 56 days before planned enrolment to reduce the number of screen failures.
* BMI ≤ 35 kg/m2
* eGFR >45 ml/min/1.73m2
* Able and willing to comply with the study protocol for the duration of the study
* Written informed consent must be obtained before any study-related assessment is performed.

Exclusion Criteria:

* Diagnosis or history indicative of monogenic, Type 2 or post-pancreatectomy diabetes
* History of >1 episode of severe (level 3) hypoglycemia in the prior 6 months
* Significant cardiovascular history defined as:

  1. History of myocardial infarction, coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accidents within six months prior to entry into the study
  2. Congestive heart failure defined as New York Heart Association (NYHA) stage III and IV
  3. Uncontrolled hypertension defined as SBP > 160 mmHg and/or DBP > 100 mmHg
  4. Symptomatic postural hypotension
  5. Use of systemic corticosteroids (except physiologic replacement doses for adrenal insufficiency) or other medications that would influence insulin sensitivity
  6. Use of non-insulin antihyperglycemic agents within prior 30 days.
  7. History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, or urological disorder including previous solid organ or cell transplant that would impact patient safety or data interpretation.
  8. History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years before screening (any history of treated cervical intraepithelial neoplasia is allowed)
  9. Known recreational substance use or psychiatric illness that, in the opinion of the Investigator, may impact the safety of the subject or objectives with scheduled visits
  10. A history of alcohol or drug abuse or drug addiction in the previous 12 months
  11. A positive pregnancy blood test for women of childbearing age or breast-feeding women 12 Are unwilling to use an "effective" method of contraception during the course of the study. Sexually active male patients, who could have children, are required to use a condom or abstained from intercourse, and refrain from sperm donation for the purposes of conception. Females have to be surgically sterile (via hysterectomy or bilateral tubal ligation) or post-menopausal or using a medically acceptable barrier method of contraception (i.e. IUD, barrier methods with spermicide or abstinence).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in AUC C-peptide | Days 0 and 84
  C-peptide level as it relates to MTX228 doses
  Change in postprandial C-peptide level area under the curve (AUC), in a 2-hour Mixed Meal Tolerance Test (MMTT), between Days 0 and 84, as well as a change in AUC C-peptide between subjects receiving different doses of MTX228.
  Justification being that the ideal dose of MTX228 will cause the largest relative increase in C-peptide levels.
Dose selection for phase IIb study | Days 0 and 84
  A change in AUC C-peptide between subjects receiving different doses of MTX228 will determine the best doses
  Justification being that the ideal dose of MTX228 will cause the largest relative increase in C-peptide levels.

SECONDARY OUTCOMES:
Lowered or increased total daily insulin dose | Days 84 and 168
  Changes in total daily insulin dose will be monitored as per:
  •Change in daily insulin use as recorded in subject's journal
  To observe if an increase in MTX228 will decrease daily insulin usage
To assess the time spent in a plasma glucose range of 3.9-10.0 mol/L | Days 84 and 168
  Changes in total daily insulin dose will be monitored based upon continuous glucose monitoring (CGM) Which dose of MTX228 helps facilitate a longer period of time spent in this optimal plasma glucose range
Time spent in high range (10.1-13.9 mmol/L) and very high range (>13.9) based upon CGM in the last two weeks of the main treatment period and separately of the extended treatment | Days 84 and 168
  Changes in total daily insulin dose will be monitored based on continuous glucose monitoring (CGM)
  Assessing which dose of MTX228 is least effective at keeping the participant out of the high and very high range. This will help aide in the dose selection phase
Change in HbA1c | Days 84 and 168
  Changes in total daily insulin dose will be monitored as per CGM and blood tests.
  Ideally, HbA1c should be lowered over time with an increased dose of MTX228
Change in fasting plasma glucose (FPG) | Days 84 and 168
  If the beneficial metabolic effects are mediated by an expansion of beta cell mass they should persist during the washout period.
The number of episodes of level 2 and 3 hypoglycemia in study participants | Days 84 and 168
  The number and duration of level 2 and 3 hypoglycemic events based upon CGM throughout treatment and follow up. Ideal doses of MTX228 should decrease the number of episodes for participants.

OTHER OUTCOMES:
Changes in AUC C-peptide between days 0 and 168, and between Days 84 and 168 in those completing the optional extension study. | days 0 and 168, and between Days 84 and 168
  •Changes observed in C-peptide or metabolic responses which increase during the extension period would support a longer treatment duration.
•Changes in secondary end-points between days 0 and 168, and between Days 84 and 168 (in subjects completing the extension study) | days 0 and 168, and between Days 84 and 168
  •Early onset type 1 diabetes is associated with a more rapid decline in beta cell mass
•Stratified analysis by baseline C-peptide level, diabetes duration, age of diabetes onset, HbA1c | days 0 and 168, and between Days 84 and 168
  The potential for beta cell regeneration may be dependent on how many beta cells are present and current metabolic demands

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada